CLINICAL TRIAL: NCT03583970
Title: Veno-arterial Extracorporeal Membrane Oxygenation Support Prior to Left Ventricular Assist Device Implantation : Initial Patients Characteristics and 6 Month Follow-up, a Retrospective Study (2013-2017) (LVAD-ECMO)
Brief Title: Veno-arterial Extracorporeal Membrane Oxygenation Prior to Left Ventricular Assist Device Implantation.
Acronym: LVAD-ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Caroline FRITZ, MD, Central Hospital, Nancy, France
Other Study IDs: PSS2017/LVADECMO-FRITZ/YB
Record Dates: First submitted 2018-06-06; First posted 2018-07-12 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Cardiogenic Shock; Heart Failure; Extracorporeal Membrane Oxygenation; Left Ventricular Assist Device
Keywords: Left Ventricular Assist Device; Extracorporeal Membrane Oxygenation; Refractory Cardiogenic Shock; Heart Failure; Cardiovascular diseases; Myocardial Infarction; Myocardial Ischemia; Shock
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure; Cardiovascular Diseases; Myocardial Infarction; Myocardial Ischemia; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Left Ventricular Assist Device Implantation — Veno-arterial extracorporeal membrane oxygenation prior to left ventricular assist device implantation : initial patients characteristics and 6 Month Follow-up

SUMMARY:
Cardiogenic shock is an uncommun pathology with a high mortatily rate around 45%. Veno arterial extracorporeal membrane oxygenation (VA-ECMO) is a temporary extracorporeal assist device which restore an adequate blood flow when a circulatory failure occures. VA-ECMO main indication is refractory cardiogenic shock whatever the etiology. Current medical care of terminal cardiac failure includes use of long-term mechanical circulatory support devices (MCSD) such as Left Ventricular Assist Device (LVAD). LVAD therapy may lead to heart transplant (bridge to transplantation), to recovery (bridge to recovery) or to permanent implantation (destination therapy). Few patients with refractory cardiogenic shock treated with VA-ECMO may secondarily need a long term MCSD with LVAD.

LVAD long-term heart assist showed interesting survival rate when implantation occured (71% after 2 years follow-up and 45% after 4 years follow-up) out of acute heart failure situation. There are only few datas concerning LVAD implantion during refractory cardiogenic shock, with a mortality between 20 to 50% in different studies.

In this way, in comparaison of current few datas on the subject of LVAD implantation under VA-ECMO, the investigators (15 french-speacking centers) would retrospectively describe a large population.

ELIGIBILITY:
Inclusion Criteria:

* Veno-arterial ExtraCorporeal Membrane Oxygenation prior to left ventricular assist device implantation.
* Veno-arterial ExtraCorporeal Membrane Oxygenation at the left ventricular assist device implantation operative time

Exclusion Criteria:

* ExtraCorporeal Membrane Oxygenation weaving before left ventricular assist device implantation.
* Cardiac assist devices other than Veno-arterial ExtraCorporeal Membrane Oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients between 01.01.2013 and 31.12.2017 in the participating centers implanted with LVAD during VA-ECMO therapy for refractory cardiogenic shock.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
6-month hospital discharge after LVAD implantation | 6 month after LVAD implantation
  6-month hospital discharge after LVAD implantation

SECONDARY OUTCOMES:
Mortality rate | up to six month after LVAD implantation
  Six month mortality rate after LVAD implantation
ICU discharge | up to six month after LVAD implantation
  Days until ICU discharge after LVAD implantation
Quality of life | up to six month after LVAD implantation
  ADL and IADL scale

OTHER OUTCOMES:
Hemodynamic Failure | Before LVAD implantation - up to 28 day - up to 6 month
  Amount of Norepinephrine infused
Cardiogenic failure | Before LVAD implantation - up to 28 day - up to 6 month
  Amount of inotrope infused
Cardio-circulatory failure | Before LVAD implantation - up to 28 day - up to 6 month
  ECLS assistance
Renal failure | Before LVAD implantation - up to 28 day - up to 6 month
  Worst KDIGO stage
Hepatic failure | Before LVAD implantation - up to 28 day - up to 6 month
  Worst values of PT/bilirubin/ AST and ALT
Thrombosis complication | Before LVAD implantation - up to 28 day - up to 6 month
  Thrombosis event
Haemorragic complication | Before LVAD implantation - up to 28 day - up to 6 month
  Haemorragic event
Respiratory failure | Before LVAD implantation - up to 28 day - up to 6 month
  Ventilation assistance
Neurological failure | Before LVAD implantation - up to 28 day - up to 6 month
  neurological sequelae
Infection complication | Before LVAD implantation - up to 28 day - up to 6 month
  documented infection

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Levy, MD-PhD, Study Chair — CHRU Nancy
Locations (1):
- CHRU Nancy, Nancy, France